CLINICAL TRIAL: NCT03552315
Title: A Randomized, Double-blind, Placebo-controlled, Crossover, Single-center, Proof of Concept Study to Evaluate the Efficacy of GoodIdea® on Glucose Homeostasis in a Healthy Population.
Brief Title: Effects of a Carbonated Water Enriched With Amino Acids and Chromium Picolinate (Good Idea®) on Glucose Homeostasis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DoubleGood AB (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DG1802
Record Dates: First submitted 2018-04-23; First posted 2018-06-11 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Postprandial Hyperglycemia; Metabolic Syndrome; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Hyperglycemia; Metabolic Syndrome; Diabetes Mellitus, Type 2 | interventions — Carbonated Water; Amino Acids; Chromium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water with amino acids and chromium (Active Comparator): The carbonated water with a proprietary blend of five amino acids and chromium picolinate is consumed with a standardized test meal to study its effects on glucose and insulin responses.
  Interventions: Dietary Supplement: Carbonated water with amino acids and chromium
- Carbonated water (Placebo Comparator): The placebo carbonated water is consumed with a standardized test meal to study its effects on glucose and insulin responses.
  Interventions: Dietary Supplement: Placebo Carbonated Water

INTERVENTIONS:
Dietary Supplement: Carbonated water with amino acids and chromium — The active carbonated water containing amino acids and chromium picolinate is consumed with a standardized test meal. Postprandial glucose and insulin response is documented for 180 minutes
  Arms: Water with amino acids and chromium
Dietary Supplement: Placebo Carbonated Water — The placebo carbonated water is consumed with a standardized test meal. Postprandial glucose and insulin response is documented for 180 minutes
  Arms: Carbonated water

SUMMARY:
It has previously been shown in healthy subjects, that a carbonated water containing a mix of amino acids and chromium picolinate can decrease postprandial blood glucose. Based on these findings, a flavored sparkling water product called Good Idea® with a proprietary blend of five amino acids and chromium picolinate has been developed. This product, along with an identical placebo, are included in this study to evaluate the effects on postprandial blood glucose in healthy, overweight adults when consumed with a standardized, high glycemic test meal. The study will be conducted in a cross-over design, double-blinded and placebo controlled, including 45 participants. The primary endpoint of the study is the incremental area under the curve (iAUC) for capillary blood glucose within 180 minutes after ingestion of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 50 years of age
* BMI 25-29.9 (±0.5) kg/m²
* Agree to maintain consistent dietary habits and physical activity levels for the duration of the study
* Healthy as determined by medical history and information provided by the volunteer
* Willingness to complete questionnaires and follow instructions associated with the study and to complete all visits
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Elevated fasting blood glucose (at or above 6.1 mmol/L)
* Women who are pregnant or breast feeding
* Any medical condition(s) or medication(s) known to significantly affect glucose metabolism. Significance to be assessed by the QI
* Use of medication, over-the-counter medication, natural health products or dietary supplements/probiotics that may affect glucose metabolism is prohibited during this study. Significance to be assessed by the qualified investigator (QI). Participants who are taking allowed prescribed medications must agree to maintain their current method and dosing regimen during the course of the study unless recommended by their physician.
* Known Type I or Type II diabetes, including women who previously have had gestational diabetes.
* Use of antibiotics within 2 weeks of enrollment
* Metabolic diseases and/or chronic gastrointestinal diseases (IBS, Crohns etc.)
* Allergy to ingredients included in investigational product, placebo or standardized meal
* Participants restricted to a vegetarian or vegan diet
* Intolerance to lactose or gluten
* Individuals who are averse to venous catheterization or capillary blood sampling
* Currently active smokers (or using other tobacco products, and e-cigarettes)
* Unstable medical conditions as determined by QI
* Participation in other clinical research trials
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Acute infection
* Any other condition which in the QI's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
The three-hour incremental area under the curve (iAUC) for capillary blood glucose, 0-180 minutes | 0, 15, 30, 45, 60, 90, 120 and 180 minutes post test meal
  The incremental area under the curve for capillary blood glucose will be measured within 180 minutes after a test meal. Blood samples will be collected at 8 time points during the 180 minutes.

SECONDARY OUTCOMES:
The three-hour iAUC for insulin, 0-180 minutes | 0, 15, 30, 45, 60, 90, 120 and 180 minutes post test meal
  The incremental area under the curve for intravenous blood insulin will be measured within 180 minutes after a test meal. Blood samples will be collected at 8 time points during the 180 minutes.
The three hour iAUC for intravenous glucose, 0-180 minutes | 0, 15, 30, 45, 60, 90, 120 and 180 minutes post test meal
  The incremental area under the curve for intravenous blood glucose will be measured within 180 minutes after a test meal. Blood samples will be collected at 8 time points during the 180 minutes.
The one-hour iAUC for intravenous Glucagon-like peptide 1 (GLP-1), 0-60 minutes | 0, 15, 30, 45 and 60 minutes post test meal
  The incremental area under the curve for intravenous blood GLP-1 will be measured within 60 minutes after a test meal. Blood samples will be collected at 5 time points during the 60 minutes.

OTHER OUTCOMES:
The three-hour Cmax of capillary blood glucose, venous blood glucose and venous blood insulin | 0, 15, 30, 45, 60, 90, 120 and 180 minutes post test meal
  Blood samples will be collected at 8 time points during the 180 minutes.
The Tmax (time to maximum concentration) of capillary blood glucose, venous blood glucose and venous blood insulin | 0, 15, 30, 45, 60, 90, 120 and 180 minutes post test meal
  Blood samples will be collected at 8 time points during the 180 minutes.
The two-hour iAUC for capillary blood glucose, venous blood glucose and venous blood insulin | 0, 15, 30, 45, 60, 90 and 120 minutes post test meal
  Blood samples will be collected at 7 time points during the 120 minutes.
The one-hour iAUC for capillary blood glucose, venous blood glucose and venous blood insulin | 0, 15, 30, 45 and 60 minutes post test meal
  Blood samples will be collected at 5 time points during the 60 minutes.
Difference in one-hour glucose (delta-glucose at 1h) from both capillary and intravenous blood. | 0 and 60 minutes post test meal
  A delta value will be calculated from samples collected at time=0 and time=60 minutes
Difference in two-hour glucose (delta-glucose at 2h) from both capillary and intravenous blood. | 0 and 120 minutes post test meal
  A delta value will be calculated from samples collected at time=0 and time=120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kristina E Andersson, PhD, Principal Investigator — Lund University and Aventure AB
Locations (1):
- Dept Experimental Medical Science, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No